CLINICAL TRIAL: NCT06482099
Title: Special Investigation for ABRYSVO Intramuscular Injection -Investigation in Pregnant Women and Infants-
Brief Title: SPECIAL INVESTIGATION FOR ABRYSVO IN PREGNANT WOMEN AND INFANTS
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3671015
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory Tract infection; RSV Vaccine; Maternal; Infant; Post Marketing Study
MeSH Terms: conditions — Respiratory Tract Infections | interventions — abrysvo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RSVpreF vaccine: Pregnant women who have been vaccinated with Abrysvo for the first time.
  Interventions: Biological: RSVpreF vaccine

INTERVENTIONS:
Biological: RSVpreF vaccine — Injection in the muscle, 1 dose 0.5mL
  Other Names: Abrysvo

SUMMARY:
This post-marketing study is a multicenter cohort study in pregnant women vaccinated with Abrysvo (RSV vaccine）designed to confirm the safety in pregnant women and their infants under actual clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who have been vaccinated with Abrysvo for the first time after Abrysvo is launched. Pregnant women who have previously participated in the clinical trials of Abrysvo will be excluded.
2. Vaccinated participants who have provided written consent regarding their participation in the study and entry of symptoms to ePRO with the use of their devices (smartphones, tablets PC, etc.) (or paper-PRO if there is any compelling reason) upon understanding the explanatory document. For a minor vaccinated participant, the parent(s) or legally acceptable representatives shall provide written consent.
3. Pregnant women who have provided written consent to the participation of their infants in the study. For a minor vaccinated participant, the parent(s) or legally acceptable representatives shall provide written consent.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who have been vaccinated with Abrysvo for the first time and their infants.
Sampling Method: Probability Sample
Enrollment: 497 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of pregnant women reporting Adverse Reactions for 28 days after vaccination | up to 28 days after vaccination
Percentage of pregnant women reporting Serious Adverse Reactions from the day of vaccination up to 28 days after delivery | up to 28 days after delivery
Percentage of pregnant women reporting reactogenicity events (local reactions and systemic events) from day of vaccination up to 7 days after vaccination | up to 7 days after vaccination
Percentage of infants reporting Adverse Reactions from the birthday up to 28 days after birth | up to 28 days after birth
Percentage of infants reporting Serious Adverse Reactions from the birthday up to 28 days after birth | up to 28 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671015